CLINICAL TRIAL: NCT04324112
Title: Phase 2 Trial of Encorafenib Plus Binimetinib for Patients With BRAF V600 Mutated Relapsed/Refractory HCL
Brief Title: Encorafenib Plus Binimetinib for People With BRAF V600 Mutated Relapsed/Refractory HCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200076; 20-C-0076
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11-06

CONDITIONS: Hairy Cell Leukemia
Keywords: MEK162; MEK1; Inhibitor; MEK2
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — binimetinib; encorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1/Experimental therapy (Experimental): Treatment with encorafenib and binimetinib
  Interventions: Drug: binimetinib; Drug: Encorafenib

INTERVENTIONS:
Drug: binimetinib — Binimetinib will be given orally at a dose of 45mg BID continuously for 28-day cycles with no resting period between cycles.
Drug: Encorafenib — Encorafenib will be given orally at a dose of 450mg QD continuously for 28-day cycles with no resting period between cycles.

SUMMARY:
Background:

Hairy cell leukemia (HCL) does not usually respond to chemotherapy. Most people with HCL have a BRAF gene mutation. This can increase the growth of cancer cells. Vemurafenib has been tested to treat these people. However, researchers think a combination of drugs might work better.

Objective:

To test if treatment with a combination of encorafenib and binimetinib in BRAF mutant

HCL is more effective than treatment with vemurafenib.

Eligibility:

People ages 18 and older with BRAF mutant HCL that did not respond to or came back after treatment

Design:

Participants will be screened with:

Medical history

Physical exam

Bone marrow biopsy: A needle will be injected through the participant s skin and into a bone to remove liquid.

Blood and urine tests

Heart and lung function tests

CT or MRI scan: Participants will lie in a machine that takes pictures of the body. They may have a contrast agent injected into a vein.

Eye exam

Participants will take the study drugs by mouth in 28-day cycles. They will take encorafenib daily. They will take binimetinib twice daily. They will keep a pill diary.

Participants will take their temperature daily.

Participants will have at least 1 visit before each cycle. Visits will include repeats of some screening tests. They will also include abdominal ultrasounds, exercise stress tests, and skin evaluations.

Participants may continue treatment as long as their disease does not get worse and they do not have bad side effects.

About a month after their last dose of treatment, participants will have a follow-up visit. Then they will have annual follow-ups....

DETAILED DESCRIPTION:
Background:

* Hairy cell leukemia (HCL) is an indolent B-cell leukemia comprising 2% of all leukemias, or approximately 1300 new cases/year in the US. The nucleoside analogs cladribine and pentostatin are highly active as monotherapy with complete remission (CR) rates of 80 to 90%. However, there is no cure from chemotherapy and patients eventually relapse with worse efficacy and cumulative toxicity (stem cell damage and neuropathy) with each repeated chemotherapy course.
* About 90% of classic HCL patients have the BRAF V600E mutation, which leads to Ras-independent activation of the MAPK pathway, causing increased phosphorylation (hyper-activation) of MEK, followed by ERK, therefore promoting the proliferation and survival of HCL cells.
* The BRAF inhibitor, vemurafenib, when used as a single agent for the treatment of HCL achieved high response rate with CR rate of 38% in 50 patients reported from 2 trials, however, treatment was limited to several months and responses lacked durability, with median CR duration of 19 months in 1 trial. In this trial, 100% of the CRs were positive for minimal residual disease (MRD) by immunohistochemistry (IHC), and failure to eradicate MRD after several months of vemurafenib likely lead to the lack of CR durability.
* In a recent trial of combined inhibition of BRAF and MEK using dabrafenib and trametinib treatment, 49% of 41 evaluable patients achieved CR, and MRD was eradicated in 15% of patients on this trial. At NIH, we enrolled a total of 28 HCL patients on this trial and achieved a CR rate of 68% amongst our patients by managing toxicity and allowing patients to remain on treatment.
* A major challenge in the long-term treatment of HCL patients with dabrafenib and trametinib is managing fever, which has necessitated long-term or intermittent steroids use for most patients.
* In the COLOMBUS trial, the combination of the BRAF inhibitor, encorafenib and the MEK inhibitor, binimetinib was found to be superior to vemurafenib for BRAF V600E+ melanoma with respect to PFS and OS and was well tolerated with low rates of toxicities including pyrexia.
* To our knowledge, neither encorafenib nor binimetinib has been tested in HCL, but the low rate of pyrexia with encorafenib plus binimetinib in melanoma suggests that this combination may be well tolerated in HCL.

Objective:

- To determine if treatment with combination encorafenib and binimetinib in BRAF V600 mutant + HCL is associated with a CR rate which exceeds that of vemurafenib.

Eligibility:

* BRAF V600 mutant HCL with at least 1 prior purine analog treatment
* Need for treatment, as evidenced by any one of the following: ANC <1 x10^3/mcL, Hgb <10g/dL, Platelet count <100 x10^3/mcL, leukemia cell count >5 x10^3/mcL, symptomatic splenomegaly, enlarging HCL mass > 2cm (>0.5cm if in central nervous system [CNS]) in short axis
* Greater than or equal to 18 years of age
* No uncontrolled infection, cardiopulmonary dysfunction, or secondary malignancy requiring treatment.
* No chemotherapy, immunotherapy, investigational agent or radiotherapy within 4 weeks prior to the start of study treatment.

Design:

* Phase 2 trial, single arm, non-randomized trial to determine if the combination of encorafenib and binimetinib achieves a CR rate in HCL which is historically higher than that of vemurafenib.
* Simon optimal 2-phase design will be used to rule out an unacceptable CR rate of 35% in favor of an improved 55% CR rate.
* Initially 12 evaluable participants will be enrolled. If 5 or more achieve CR, then accrual will continue to a total of 32 evaluable participants
* Encorafenib will be given at a dose of 450mg QD and binimetinib at a dose of 45mg BID for as long as participants can continue dosing chronically without significant toxicity or a trial off therapy due to achievement of MRD negative complete remission or PR/CR in which they would like a trial off therapy. Participants may return to therapy within 2 years of stopping treatment if evidence of disease returns.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically confirmed diagnosis of HCL according to morphological and immunophenotypic criteria of World Health Organization (WHO) classification [WHO, 2008 revised 2016] of lymphoid neoplasm. Participants should have at least one of the following indications for therapy:

  * Absolute neutrophil count (ANC) <1 x10(3)/mcL
  * Hemoglobin <10g/dL
  * Platelets<100 x10(3)/mcL
  * Symptomatic splenomegaly
  * Enlarging HCL mass > 2cm in short axis (>0.5cm in short axis for CNS mass)
  * Leukemia cell count>5x10(3)/mcL

Participants who have eligible blood counts within 4 weeks prior to initiation of study therapy will not be considered ineligible if subsequent blood counts prior to initiation of study therapy fluctuate and become ineligible up until the time of the initiation of study therapy.

* Participants must have BRAF V600 mutation as confirmed from fresh bone marrow aspirate, peripheral blood sample, or lymph node/mass by the Laboratory of Pathology, NCI. This may be done by PCR or sequence-based assays.
* Participants who are ineligible for, unable to obtain in a timely manner, cannot access, unwilling to undergo or have failed Moxetumomab Pasudotox trial at NCI
* Refractory or relapsed disease- defined as either:

  * Refractory- no response or disease progression in <=1 year following first-line treatment with a purine analog, or
  * Relapsed- having relapsed following treatment with at least 1 prior purine-analog treatment
* Age >=18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <=2 (Karnofsky >=60%)
* Participants must have adequate organ and marrow function as defined below:

  * Total bilirubin <= 3x upper limit of normal (ULN), unless consistent with Gilbert s (ratio between total and direct bilirubin > 5)
  * AST and ALT <= 3x ULN
  * Alkaline phosphatase < 2.5x ULN
  * Serum creatinine <= 1.5 mg/dL or creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal calculated using estimated glomerular filtration rate (eGFR)
  * Serum albumin >= 2 g/dL
  * Prothrombin time (PT)/International Normalized Ratio (INR) < 2.5x ULN (If on warfarin, PT/INR < 3.5x ULN; If on any other anticoagulation, (PT) < 2.5x ULN
  * Fibrinogen >= 0.5x lower limit of normal
  * Females of childbearing potential (FOCBP) who are sexually active with a non-sterilized male partner must use a highly effective method of contraception and not donate ova prior to study entry and or the duration of study treatment and until 30 days after the last dose of study drug. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. There is a potential for encorafenib to induce CYP3A4, which may reduce the effectiveness of hormonal contraception methods. Therefore, the use of at least 1 form of non-hormonal contraception is required for females of childbearing potential during study

treatment in this study. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or those who are premenarchal or postmenopausal (defined as 12 months with no menses without an alternative medical cause). A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Not all methods of contraception are highly effective. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

--Male participants must use a condom during treatment and through 90 days after the end of systemic exposure to study drug/treatment. If the male participant has a partner that is of child-bearing potential, the partner should also use contraception through

90 days after the end of systemic exposure to study drug/treatment. In addition, male participants must refrain from donating sperm during the study treatment and through 90 days after the end of systemic exposure to study drug/treatment. Males who have had a vasectomy qualify as having met the requirement for a highly effective birth control method.

* Nursing participants must be willing to discontinue nursing from study treatment initiation through 14 days after the last dose of the study drugs.
* Ability of participant to understand and the willingness to sign a written informed consent document.
* Must co-enroll in study 10-C-0066: Collection of Human Samples to Study Hairy Cell and other Leukemias, and to Develop Recombinant Immunotoxins for Cancer Treatment

EXCLUSION CRITERIA:

* Participants who have had chemotherapy, immunotherapy, investigational agent or radiotherapy within 4 weeks prior to the start of study treatment.
* Prior therapy with encorafenib and/or binimetinib
* Participants who are receiving any other investigational agents or have received an investigational agent within 14 days prior to the start of study treatment.
* Participants who have undergone major surgery <=6 weeks prior to start of study treatment or who have not recovered from side effects of such procedure
* Known hypersensitivity or contraindication to any component of binimetinib or encorafenib or their excipients
* Inability to swallow and retain study drugs.
* Pregnant women as evaluated by a positive serum or urine beta-human chorionic gonadotropin (beta-hCG).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiac dysfunction, uncontrolled pulmonary infection, pulmonary edema or psychiatric illness/social situations that would limit compliance with study requirements.
* Evidence of active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection. Note: Participants with laboratory evidence of cleared HBV or HCV infection may be enrolled. If positive for Hepatitis B core antibody or surface antigen the participant must be on Tenofovir or Entecavir and Hepatitis B deoxyribonucleic acid (DNA) viral load must be <2000 IU/mL
* Active second malignancy requiring treatment other than minor resection of indolent cancers like basal cell and squamous skin cancers.
* Human immunodeficiency virus (HIV)-positive participants unless taking appropriate anti-HIV medications with a CD4 count of > 200. Otherwise, there may be an increased risk of infections.
* History of an allogeneic bone marrow or stem cell transplant.
* Known history of chronic pancreatitis.
* Impaired cardiovascular function or clinically significant cardiovascular disease including, but not limited to, any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) <3months prior to initiation of study therapy
  * Congestive heart failure requiring treatment (New York Heart Association Grade greater than or equal to 2);
  * Left ventricular ejection fraction (LVEF) < 50% as determined by Multigated Acquisition Scan (MUGA) or Transthoracic echocardiogram (TTE);
  * Uncontrolled hypertension defined as persistent systolic blood pressure greater than or equal to 160 mmHg or diastolic blood pressure greater than or equal to 100 mmHg despite current therapy;
  * History or presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia);
  * Triplicate average baseline QTcF interval greater than or equal to 480 ms.
* Impairment of gastrointestinal function or disease which may significantly alter the absorption of study drug (e.g., active ulcerative disease, uncontrolled vomiting or diarrhea, malabsorption syndrome, small bowel resection with decreased intestinal

absorption), or recent (less than or equal to 3 months) history of a partial or complete bowel obstruction, or other conditions that will interfere significantly with the absorption of oral drugs.

* Concurrent neuromuscular disorder that is associated with elevated creatinine kinase CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of maculopathy or retinopathy for which there is an increased risk

of MEK induced exudation (e.g., Central Serous Retinopathy).

* History of thromboembolic or cerebrovascular events less than or equal to 12 weeks prior to the first dose of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli.
* Note: Participants with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for at least 4 weeks.
* Note: Participants with thromboembolic events related to indwelling catheters or other procedures may be enrolled
* Participants taking strong CYP3A4 inhibitors and strong/moderate CYP3A4 inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
CR rate | every year
  determine if treatment with combination encorafenib and binimetinib in BRAF V600 mutant + HCL is associated with a CR rate which exceeds that of vemurafenib

SECONDARY OUTCOMES:
MRD negative CR | every year
  Fraction of patients who achieve MRD negative CR after treatment with encorafenib and binimetinib
time to next treatment | every year
  duration of time from the start of the study drugs to next line of treatment
overall survival | every year
  the time from the start of the treatment until time of death from any cause
event free survival | every year
  the time from study enrollment to the first occurrence of progression, relapse after response, or death from any cause
duration of response | every year
  the time criteria are met for CR or PR (whichever is recorded first) until the first date that patient no longer qualifies as a PR
progression free-survival | every year
  duration of time from the start of the treatment until time of disease relapse from PR, disease progression, or death, whichever occurs first
rate of pyrexia | every year
  fraction of patients that have pyrexia at any time while on study

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0076.html